CLINICAL TRIAL: NCT04953104
Title: A Phase II Clinical Trial to Investigate ARID1A and/or KDM6A Mutation and CXCL13 Expression in the Pre-treatment Tumor Samples as a Combinatorial Predictive Biomarker for Immune Checkpoint Therapy in Metastatic Urothelial Cancer
Brief Title: ARID1A and/or KDM6A Mutation and CXCL13 Expression
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0104; NCI-2021-05785 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0104 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Bladder Urothelial Carcinoma; Locally Advanced Renal Pelvis Urothelial Carcinoma; Locally Advanced Ureter Urothelial Carcinoma; Locally Advanced Urethral Urothelial Carcinoma; Locally Advanced Urothelial Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis Urothelial Carcinoma; Metastatic Ureter Urothelial Carcinoma; Metastatic Urethral Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Recurrent Bladder Urothelial Carcinoma; Recurrent Renal Pelvis Urothelial Carcinoma; Recurrent Ureter Urothelial Carcinoma; Recurrent Urethral Urothelial Carcinoma; Recurrent Urothelial Carcinoma; Stage III Bladder Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage III Urethral Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8; Stage IIIB Bladder Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Renal Pelvis Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8; Stage IVA Bladder Cancer AJCC v8; Stage IVB Bladder Cancer AJCC v8; Unresectable Bladder Urothelial Carcinoma; Unresectable Renal Pelvis Urothelial Carcinoma; Unresectable Ureter Urothelial Carcinoma; Unresectable Urethral Urothelial Carcinoma; Unresectable Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — Nivolumab; relatlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab & relatlimab) (Experimental): Participants found to be eligible to take part in this study, you will receive nivolumab and relatlimab by vein over about 30 minutes on Day 1 of every 28-day study cycle (about every 4 weeks).
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Biological: Nivolumab; Drug: Relatlimab

INTERVENTIONS:
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Drug: Relatlimab — Given IV
  Other Names: BMS-986016

SUMMARY:
This phase II trial studies the effect of nivolumab in urothelial cancer that has spread to other places in the body (metastatic), specifically in patients with aberrations in ARID1A gene (ARID1A mutation) and correlate with expression level of CXCL13, an immune cytokine. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving nivolumab may help control the disease in patients with urothelial cancer or solid tumors. This trial aims at enriching patient selection based on genomic and immunological attributes of the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate objective response rate (ORR) and overall survival (OS) in participants with ARID1A and/or KDM6A mutations receiving nivolumab and relatlimab combination therapy. II. To estimate objective response rate (ORR) and overall survival (OS) in participants with ARID1A and/or KDM6A mutations plus CXCL13-high expression and ARID1A and/or KDM6A mutations plus CXCL13-low expression, receiving nivolumab and relatlimab therapy.

SECONDARY OBJECTIVES:

I. To estimate progression free survival (PFS) in subjects with harboring ARID1A and/or KDM6A mutation treated with nivolumab and relatlimab combination therapy.

II. To estimate progression free survival (PFS) in subjects with ARID1A and/or KDM6A mutations plus CXCL13-high expression and ARID1A and/or KDM6A mutations plus CXCL13-low expression, treated with nivolumab and relatlimab combination therapy.

III. To assess peripheral and tumor infiltrating immune cell sub-populations in patients with ARID1A mutations, KDM6A mutations, ARID1A plus CXCL13-high and ARID1A plus CXCL13-low expression, KDM6A plus CXCL13-high and KDM6A plus CXCL13-low expression, to determine predictors of response and resistance.

IV. To determine the expression pattern of CXCL13 in ARID1A and/or KDM6A mutant tumors

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Cycles repeats 28 days (4 weeks) for up to 2 years in the absence of disease or unacceptable toxicity.

After the completion of study treatment, patients are followed up for 100 days, then every 3-6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will have a tumor harboring genomic mutation of ARID1A and/or KDM6A. ARID1A and/or KDM6A mutation testing will be performed as standard of care.
2. Histological or cytological evidence of metastatic or surgically unresectable urothelial cell carcinoma of the urothelial involving the bladder, urethra, ureter, or renal pelvis. Minor histologic variants (< 50% overall) are acceptable.
3. Participants must have progression or recurrence after treatment i) with at least 1 platinum-containing chemotherapy regimen for metastatic or surgically unresectable locally advanced urothelial cancer, or ii) are ineligible or refused frontline chemotherapy.
4. All participants must have measurable disease by CT or MRI per RECIST 1.1 criteria.
5. Evaluable tumor tissue (archived or new biopsy) must be provided for biomarker analysis as FFPE tumor block or minimum of 10 slides. Archived tissue may be from prior biopsy of unresectable or metastatic disease or from prior surgical resection. Request for available archival tissue must be in process prior to registration.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
7. Prior palliative radiotherapy must have been completed at least 2 weeks prior to study drug administration. Participants with progression in a previously radiated field will also be eligible.
8. Screening laboratory values must meet the following criteria and must be obtained within 7 days prior to first dose:

   i. Neutrophils ≥ 1000/µL ii. Platelets ≥ 100 x1 x103/µL iii. Hemoglobin ≥ 8.0 g/dL iv. AST and ALT ≤ 3 x ULN (or ≤ 5 X ULN for participants with liver metastases).

   v. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) vi. Serum creatinine ≤ 2 x ULN or creatinine clearance (CrCl) ≥ 30 mL/min (using the

   Cockcroft-Gault formula):

   Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL vii. Troponin T (TnT) or I (TnI) ≤ 2 x institutional ULN. Participants with TnT or TnI levels between > 1 to 2 × ULN will be permitted if a repeat levels within 24 hours are

   ≤ ULN. If TnT or TnI levels are between > 1 to 2 × ULN within 24 hours, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 × ULN, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation.

   viii. Re-enrollment: This study permits the re-enrollment of a participant that has discontinued the study as a pre-treatment failure (ie, subject has not been treated). If re-enrolled, the participant must be re-consented and inclusion/exclusion criteria reassessed.
9. Participants are required to participate in PA13-0291 for correlative studies. Participants will need to consent for biopsy and peripheral blood collection as documented in the study calendar.
10. Females of childbearing potential (FCBP) must agree to follow instructions for method(s) of contraception from the time of enrollment, for the duration of study treatment, and for 5 months after the last study dose of study treatment (see Section 8.5).
11. Males who are sexually active with FCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment (see Section 8.5). Male participants should refrain from donating sperm during the study.
12. FCBP must have a negative serum or urine pregnancy test within 24 hours prior to the start of study treatment.

Exclusion Criteria:

1. Prior treatment with an anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
2. Active brain metastases or leptomeningeal metastases. Participants with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment is complete and within 14 days prior to first dose of study drug administration. Where MRI is contraindicated CT scan is acceptable. Cases must be discussed with the medical monitor. Brain lesions are not considered measurable disease. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
3. Any serious or uncontrolled medical disorder, that in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the participant to receive protocol therapy, or interfere with the interpretation of study results.
4. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, prostate cancer without evidence of PSA progression or carcinoma in situ such as the following: gastric, prostate, cervix, colon, melanoma, or breast for example.
5. Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism, due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
6. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
7. All toxicities attributed to prior anti-cancer therapy other than neuropathy, alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 5) or baseline before administration of study drug. Participants with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll. Neuropathy must have resolved to Grade 2 (NCI CTCAE version 5).
8. Treatment with any chemotherapy, radiation therapy, biologics for cancer, or investigational therapy within 14 days or five (5) half-lives whichever is shorter, of first administration of study treatment. Prior palliative radiotherapy must have been completed at least 2 weeks prior to study drug administration as indicated in inclusion criteria h.
9. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (RNA) or hepatitis C antibody (HCV antibody) indicating acute or chronic infection.
10. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  Defined as the rate of confirmed complete responses + partial responses as determined by Response Evaluation Criteria in Solid Tumors 1.1 criteria and as assessed by the investigator. In addition, will also calculate the posterior probability that ORR is bigger in CXCL13 high group than in the CXCL low group.
Overall survival (OS) | From date of first study treatment to death due to any cause, assessed up to 2 years
  The Kaplan-Meier method will be used to estimate the median OS and 1-year survival rate; the 95% confidence interval (CI) of the 1-year survival rate will also be reported.

OTHER OUTCOMES:
Progression free survival (PFS) | Up to 2 years
  Will be estimated using the Kaplan-Meier method and compared using the log rank test. Cox proportional Hazard models will be used to evaluate the association between PFS or OS and ARID1A mutation / CXCL13 expressions to evaluate their utility as predictive biomarkers for efficacy.
  Logistic regression models will be fitted to explore the association between response and ARID1A mutation / CXCL13 expressions to evaluate their utility as predictive biomarkers for efficacy.
Overall survival | Up to 2 years
  Will be estimated using the Kaplan-Meier method and compared using the log rank test. Cox proportional Hazard models will be used to evaluate the association between PFS or OS and ARID1A mutation / CXCL13 expressions to evaluate their utility as predictive biomarkers for efficacy.
  Logistic regression models will be fitted to explore the association between response and ARID1A mutation / CXCL13 expressions to evaluate their utility as predictive biomarkers for efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Goswami, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org